CLINICAL TRIAL: NCT02372188
Title: Effect of Caffeine With and Without a Bitter Masking Compound on Gastric pH, Taking Into Account the Effect on Satiety Hormones in Blood Plasma and on Food Intake
Brief Title: Influence of a Bitter Compound and Bittermasking Compound on Gastric pH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Veronika Somoza, Univ.-Prof. Dr., University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GAS-14
Record Dates: First submitted 2014-12-19; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Change of Gastric pH
MeSH Terms: interventions — Water; Caffeine

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Water (Experimental): 125 mL water are administered during or before gastric pH measurement
  Interventions: Other: water
- Caffeine (Experimental): 150 mg Caffeine and 125 mL water are administered during or before gastric pH measurement
  Interventions: Dietary Supplement: caffeine
- Caffeine + homoeriodictyol sodium salt (Experimental): 150 mg Caffeine + 30 mg homoeriodictyol sodium salt and 125 mL water are administered during or before gastric pH measurement
  Interventions: Dietary Supplement: caffein + homoeriodictyol sodium salt
- homoeriodictyol sodium salt (Experimental): 30 mg homoeriodictyol sodium salt and 125 mL water are administered during the gastric pH measurement
  Interventions: Dietary Supplement: homoeriodictyol sodium salt

INTERVENTIONS:
Other: water — Control
  Arms: Water
Dietary Supplement: caffeine
  Arms: Caffeine
Dietary Supplement: caffein + homoeriodictyol sodium salt
  Arms: Caffeine + homoeriodictyol sodium salt
Dietary Supplement: homoeriodictyol sodium salt
  Arms: homoeriodictyol sodium salt

SUMMARY:
The purpose of this study is to elucidate whether bitter taste induced by the bitter compound caffeine and the reduction of bitter taste by addition of the bitter masking compound Homoeriodictyol sodium salt (HED) influence gastric acid secretion, subjective feelings of hunger, ad libitum food intake and satiating hormones in healthy volunteers.

DETAILED DESCRIPTION:
The influence of 125 mL water, 150 mg caffeine/125 mL water, 30 mg HED/125 mL water or the combination of 150 mg caffeine + 30 mg HED/125 mL water on the gastric pH on different test days was investigated. Prior to the intervention, the trial subjects had to fast from food and liquid for 10 h, except for 200 mL of tap water that were allowed during this time period. During the experiment, the subjects remained in a supine left-sided position.

For the non-invasive measurement of the gastric pH, the Heidelberg Detection System (Heidelberg Medical Inc., USA) was used which has been successfully used in our working group.

This system consists of a pH-sensitive capsule (called a Heidelberg capsule), with a length of 2 cm, that has to be swallowed and contains a miniature radio transmitter. This system allows the detection of the actual gastric pH of the volunteer over a specific time period [Liszt et al 2012, Rubach et al. 2014].

Prior to each test, Heidelberg capsules were activated for 5 min in a 0.9% sterile NaCl solution and calibrated using two calibration points, pH 1 and 7. Afterward, the subjects swallowed the capsule lay down on the left side. The capsule sends a signal to a transceiver, which has to be placed on the abdomen of the volunteer. The transceiver sends the signal to the recorder connected to a computer. The data can be collected and shown as a gastrogram on the computer screen, where the pH is drawn over time. When the intragastric pH was constant between pH 0.5 and 2.5 for at least 3 min, the capsule was considered to be in the stomach. Afterward, each trial started with the administration of 5 mL of a saturated sodium bicarbonate solution (NaHCO3). This alkaline challenge triggers a rise in gastric pH between around pH 6 to 7 and subsequently leads to the secretion of stomach acid by the parietal cells. The test solutions were administered 5 minutes after or 30 min before the alkaline challenge.

Reacidification time as well as the time until start of the reacidification has been analyzed.

Ratings of hunger were assessed before and after each gastric pH measurement by means of visual analog scales (VAS). Before and after each intervention blood samples were drawn to quantify satiety hormones (ghrelin, PYY, GLP-1, serotonin). Ad libitum energy and macronutrient intakes from a standardized breakfast served after each treatment were calculated.

ELIGIBILITY:
Inclusion Criteria:

* good general state of health
* sensorically untrained
* BMI: 19 - 26 kg/m2

Exclusion Criteria:

* gastro-intestinal disease or discomfort,
* metabolic diseases,
* H.pylori infection,
* smoking,
* increased sensibility towards caffeine,
* intake of antibiotics in the last 2 months,
* medication except for oral contraceptives,
* drug- or alcohol-abuse,
* heart disease, high blood pressure,
* pregnancy

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Change of the intragastral pH determined by the Heidelberg Detection system | recorded over a time period from 1 - 60 min

SECONDARY OUTCOMES:
Change of plasma levels of Serotonin, Ghrelin, PYY and GLP-1 | Plasma are taken at two time points before and after the gastric pH measurement during a time period between 15 - 60 min
  higher plasma levels of serotonin, PYY and GLP-1 are a satiety signal while higher levels of Ghrelin, Hunger-stimulating hormone, indicate appetite
Food intake | after the gastric pH measurement on each testing day the subjects are served an ad libitum breakfast, and they have an open time frame how long they want to eat, max. 1 hour is anticipated
  A weighed standard breakfast will be served and ad libitum energy intake will be assessed by weighing the left overs of the breakfast and analyzed by nutrient data base. Total caloric intake [kcal], as well as the total carbohydrate [g], protein [g] and fat [g] intake will be analyzed.
subjective feelings of hunger are recorded by means of visual analog scales (VAS) | subjects are asked to fill the VAS out immediately before and after the gastric pH measurement, max. 2 min is anticipated
  The volunteers have to make a sign on a 10 cm long scale (visual analog scale), ranging from 0 (not hungry) to 10 (very hungry). The volunteer can make the sign at any point of the scale and we will measure the distance from the beginning until the sign [cm].

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Somoza, Prof. PhD, Principal Investigator — University of Vienna
Locations (1):
- Christian Doppler Laboratory for Bioactive Aroma Compounds, Vienna, Austria

REFERENCES:
- [Background] Liszt KI, Walker J, Somoza V. Identification of organic acids in wine that stimulate mechanisms of gastric acid secretion. J Agric Food Chem. 2012 Jul 18;60(28):7022-30. doi: 10.1021/jf301941u. Epub 2012 Jul 5. PMID 22708700
- [Background] Rubach M, Lang R, Bytof G, Stiebitz H, Lantz I, Hofmann T, Somoza V. A dark brown roast coffee blend is less effective at stimulating gastric acid secretion in healthy volunteers compared to a medium roast market blend. Mol Nutr Food Res. 2014 Jun;58(6):1370-3. doi: 10.1002/mnfr.201300890. Epub 2014 Feb 8. PMID 24510512